CLINICAL TRIAL: NCT01178125
Title: A Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of a Combination Oral Contraceptive Regimen (DR-102) for the Prevention of Pregnancy in Women
Brief Title: A Study to Evaluate the Efficacy and Safety of DR-102 for the Prevention of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DSG-PPS-303
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Contraception; Female Contraception
Keywords: Pregnancy Prevention; Oral Contraceptives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DR-102 (Experimental): desogestrel/ethinyl estradiol 0.15/0.02 mg for 21 days then ethinyl estradiol 0.01 mg for 7 days
  Interventions: Drug: DR-102

INTERVENTIONS:
Drug: DR-102

SUMMARY:
This is an open-label, single treatment study. All subjects will receive 12 months of oral contraceptive therapy with DR-102. Study participants will receive physical and gynecological exams, including Pap smear. During the study, all participants will be required to complete a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active at risk for pregnancy
* Agreement to use study oral contraceptive therapy as their only method of birth control during the study
* History of regular spontaneous menstrual cycles or withdrawal bleeding episodes
* Others as dictated by protocol

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Pregnancy or plans to become pregnant in the next 14 months
* Smoker and age greater than or equal to 35 years
* Others as dictated by protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2858 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Women's Health Research Protocol Chair, Study Chair — Teva Women's Health
Locations (62):
- United States (52):
  - Teva Investigational Site 10007, Montgomery, Alabama
  - Teva Investigational Site 10013, Phoenix, Arizona
  - Teva Investigational Site 10017, Phoenix, Arizona
  - Teva Investigational Site 10032, Little Rock, Arkansas
  - Teva Investigational Site 10026, San Diego, California
  - Teva Investigational Site 10056, San Diego, California
  - Teva Investigational Site 10002, Colorado Springs, Colorado
  - Teva Investigational Site 10033, Colorado Springs, Colorado
  - Teva Investigational Site 10057, Washington D.C., District of Columbia
  - Teva Investigational Site 10052, Clearwater, Florida
  - Teva Investigational Site 10021, Jacksonville, Florida
  - Teva Investigational Site 10036, Leesburg, Florida
  - Teva Investigational Site 10012, Miami, Florida
  - Teva Investigational Site 10015, Miami, Florida
  - Teva Investigational Site 10055, Palm Beach Gardens, Florida
  - Teva Investigational Site 10001, West Palm Beach, Florida
  - Teva Investigational Site 10031, Decatur, Georgia
  - Teva Investigational Site 10041, Roswell, Georgia
  - Teva Investigational Site 10050, Savannah, Georgia
  - Teva Investigational Site 10008, Louisville, Kentucky
  - Teva Investigational Site 10023, Mount Sterling, Kentucky
  - Teva Investigational Site 10048, Lawrenceville, New Jersey
  - Teva Investigational Site 10030, Moorestown, New Jersey
  - Teva Investigational Site 10014, Albuquerque, New Mexico
  - Teva Investigational Site 10006, Rochester, New York
  - Teva Investigational Site 10044, Cary, North Carolina
  - Teva Investigational Site 10040, Charlotte, North Carolina
  - Teva Investigational Site 10034, New Bern, North Carolina
  - Teva Investigational Site 10018, Winston-Salem, North Carolina
  - Teva Investigational Site 10046, Winston-Salem, North Carolina
  - Teva Investigational Site 10022, Columbus, Ohio
  - Teva Investigational Site 10039, Columbus, Ohio
  - Teva Investigational Site 10028, Oklahoma City, Oklahoma
  - Teva Investigational Site 10043, Philadelphia, Pennsylvania
  - Teva Investigational Site 10003, Pittsburgh, Pennsylvania
  - Teva Investigational Site 10049, Bluffton, South Carolina
  - Teva Investigational Site 10037, Columbia, South Carolina
  - Teva Investigational Site 10035, Greenville, South Carolina
  - Teva Investigational Site 10047, Mt. Pleasant, South Carolina
  - Teva Investigational Site 10016, Jackson, Tennessee
  - Teva Investigational Site 10045, Knoxville, Tennessee
  - Teva Investigational Site 10005, Memphis, Tennessee
  - Teva Investigational Site 10042, Nashville, Tennessee
  - Teva Investigational Site 10054, Dallas, Texas
  - Teva Investigational Site 10019, Houston, Texas
  - Teva Investigational Site 10020, San Antonio, Texas
  - Teva Investigational Site 10038, Arlington, Virginia
  - Teva Investigational Site 10024, Norfolk, Virginia
  - Teva Investigational Site 10051, Norfolk, Virginia
  - Teva Investigational Site 10053, Richmond, Virginia
  - Teva Investigational Site 10027, Seattle, Washington
  - Teva Investigational Site 10029, Tacoma, Washington
- Israel (10):
  - Teva Investigational Site 80108, Beersheba
  - Teva Investigational Site 80109, Giv‘atayim
  - Teva Investigational Site 80104, Haifa
  - Teva Investigational Site 80107, Haifa
  - Teva Investigational Site 80101, Modiin
  - Teva Investigational Site 80103, Or Yehuda
  - Teva Investigational Site 80100, Petah Tikva
  - Teva Investigational Site 80105, RishonLe'zio
  - Teva Investigational Site 80102, Tel Aviv
  - Teva Investigational Site 80106, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3691 women desiring pregnancy prevention were screened for enrollment into this study. Of the 3691 subjects screened, 2858 subjects at 53 centers in the US and 9 centers in Israel met entry criteria and were considered to be eligible for enrollment into the study.
Pre-assignment Details: Of the 2858 enrolled, 93 participants withdrew from study before taking any investigational product, for the following reasons: lost to follow-up (n=34), consent withdrawn (n=17), sponsor request (n=13), withdrawn due to pregnancy (n=11), noncompliance (n=6), other (n=6), protocol violation (n=3), adverse event(n=2), investigator request (n=2).
Period: Overall Study
Arm/Group | DR-102
Started | 2858 (Number enrolled.)
Safety Population | 2765 (Received at least 1 dose of DR-102.)
Intent to Treat (ITT) Population | 2607 (Completed at least one 28-day cycle of investigational product.)
Pregnancy ITT (PITT) Population | 2401 (Participants in the ITT population between the ages of 18 and 35, inclusive.)
Completed | 1680
Not Completed | 1178
Not completed — Lost to Follow-up | 397
Not completed — Adverse Event | 244
Not completed — Withdrawal by Subject | 209
Not completed — Noncompliance | 184
Not completed — Pregnancy | 55
Not completed — Other Reason | 39
Not completed — Sponsor Decision | 28
Not completed — Protocol Violation | 17
Not completed — Investigator Decision | 5

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | DR-102
Number analyzed (Participants) | 2765
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2765
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1798
  Black | 428
  Asian | 72
  Hispanic | 393
  Other | 74
Weight [Mean (Standard Deviation); unit: kg] — n=2764 (1 participant did not have a value recorded for weight)
  kg | 72.4 (18.62)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — n=2763 (2 participants did not have values recorded for BMI)
  kg/m^2 | 26.9 (6.54)

OUTCOME MEASURES:

1. Primary Outcome: All Users Pregnancy Rates Based on Pearl Index (PI) Analyses for 28-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight, Using the 7-Day Rule
Description: Contraceptive failure is measured by the pregnancy rate calculated using the Pearl Index (PI) and the 7-day rule (a standardized process for calculating pregnancy rates). PI used all pregnancies, as determined by a positive urine and/or serum pregnancy test, except those for which the date of conception was before starting DR-102 or > 7 days after stopping the combination desogestrel/ethinyl estradiol (DSG/EE) or ethinyl estradiol (EE) treatment of DR-102.The PI is defined as number of contraceptive failures per 100 women-years of exposure: (100)*(total number of pregnancies)*(13)/(total number of 28-day cycles). Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'All Users' set included PITT participants who completed at least one 28-day cycle.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Units Other Than Participants: Treatment Cycles
Groups:
- DR-102: Total: All participants taking desogestrel/ethinyl estradiol 0.15/0.02 mg for 21 days then ethinyl estradiol 0.01 mg for 7 days
- DR-102: Baseline Body Weight <90 kg: Subpopulation of total participants with a Baseline body weight <90 kg
- DR-102: Baseline Body Weight ≥90 kg: Subpopulation of total participants with a Baseline body weight ≥90 kg
Arm/Group | DR-102: Total | DR-102: Baseline Body Weight <90 kg | DR-102: Baseline Body Weight ≥90 kg
Number analyzed (Participants) | 2401 | 2034 | 367
Number analyzed (Treatment Cycles) | 24631 | 21050 | 3581
pregnancies / 100 woman years exposure | 2.43 [1.778 to 3.237] | 2.35 [1.661 to 3.220] | 2.90 [1.254 to 5.716]

2. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Due to AEs
Description: AEs summarized are those that began or worsened after treatment with investigational product (IP). An AE is any untoward medical occurrence in a subject or clinical investigation subject participating in a clinical study and which does not necessarily have to have a causal relationship with this treatment or clinical study. Severity of AEs was assessed as mild, moderate or severe. A severe AE was defined as incapacitating, with inability to perform usual activity. An AE was defined as treatment-related when there is reasonable possibility that the AE was caused by or attributed to the IP and/or a causal relationship cannot be ruled out. An SAE was defined as one that meets any one of the following criteria: fatal or life-threatening; requires or prolongs in-patient hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical event.
Time Frame: Serious adverse Event (SAE) reporting period began upon signed informed consent and ended at the Final Study or the Early Withdrawal Visit. AEs were reported at each study visit (Weeks 0 through Week 53). Treatment duration with IP was up to one year.
Population: Safety population (received at least 1 dose of DR-102)
Measure: Number; unit: participants
Arm/Group | DR-102
Number analyzed (Participants) | 2765
participants
  Any AE | 1778
  Severe AEs | 173
  Treatment-related AEs | 608
  Deaths | 0
  Other SAEs | 46
  Withdrawn From Study Due to AEs | 234

3. Other Pre Specified Outcome: Endometrial Biopsy Classification Results for Endometrial Tissue/Glands at Baseline and Endpoint
Description: A subset of study participants agreed to have baseline and endpoint (Week 51/Early Withdrawal) endometrial biopsies. Results were provided for assessment of endometrial tissue/glands. Atrophic: scant or moderate amount of tissue, consists of tiny strips and wisps of surface endometrium or small tubular glands with scant or absent luminal secretions. Inactive: tubular glands lined by epithelial cells with mild pseudostratified and elongated nuclei. Proliferative: tubular or elongated glands lined by cells with elongated, dense, pseudostratified nuclei. Secretory: glands are tortuous or coiled with subnuclear vacuolation, secretion, and intraluminal tufts. Hyperplasia: proliferative type of glands showing glandular crowding with irregular shapes and sizes of enlargement, budding, and branching. Menstrual: glandular and stromal breakdown with fibrin thrombi in small vessels, condensed and collapsed stroma, and necrotic debris.
Time Frame: Baseline (at Enrollment), Endpoint (Week 51/Early Withdrawal)
Population: Subset of participants with sufficient tissue at both Baseline and Endpoint biopsies.
Measure: Number; unit: participants
Groups:
- DR-102: Baseline: prior to starting desogestrel/ethinyl estradiol 0.15/0.02 mg for 21 days then ethinyl estradiol 0.01 mg for 7 days
- DR-102: Endpoint: at Week 51 of treatment with desogestrel/ethinyl estradiol 0.15/0.02 mg for 21 days then ethinyl estradiol 0.01 mg for 7 days
Arm/Group | DR-102: Baseline | DR-102: Endpoint
Number analyzed (Participants) | 72 | 72
participants
  Atrophic | 10 | 47
  Inactive | 13 | 6
  Proliferative | 11 | 9
  Secretory | 38 | 10
  Hyperplasia | 0 | 0
  Menstrual Endometrium | 0 | 0

4. Secondary Outcome: All Users Life-Table Estimates of Pregnancy Rates Based on 28-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: A life table approach was used to estimate the cumulative pregnancy rate on a cycle-by-cycle basis for each of the thirteen 28-day treatment cycles.
Time Frame: thirteen 28-day cycles
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: pregnancies / cumulative exposure
Arm/Group | DR-102: Total | DR-102: Baseline Body Weight <90 kg | DR-102: Baseline Body Weight ≥90 kg
Number analyzed (Participants) | 2401 | 2034 | 367
pregnancies / cumulative exposure
  Cycle 1 | 0.0004 [0.0001 to 0.0030] | 0.0005 [0.0001 to 0.0035] | 0 [0.0000 to 0.0000]
  Cycle 2 | 0.0013 [0.0004 to 0.0039] | 0.0010 [0.0002 to 0.0040] | 0.0028 [0.0004 to 0.0198]
  Cycle 3 | 0.0031 [0.0015 to 0.0064] | 0.0031 [0.0014 to 0.0069] | 0.0028 [0.0004 to 0.0198]
  Cycle 4 | 0.0073 [0.0045 to 0.0119] | 0.0070 [0.0041 to 0.0120] | 0.0091 [0.0029 to 0.0280]
  Cycle 5 | 0.0078 [0.0049 to 0.0125] | 0.0070 [0.0041 to 0.0120] | 0.0125 [0.0047 to 0.0330]
  Cycle 6 | 0.0088 [0.0056 to 0.0138] | 0.0082 [0.0049 to 0.0136] | 0.0125 [0.0047 to 0.0330]
  Cycle 7 | 0.0104 [0.0069 to 0.0158] | 0.0094 [0.0059 to 0.0151] | 0.0163 [0.0068 to 0.0388]
  Cycle 8 | 0.0132 [0.0091 to 0.0192] | 0.0120 [0.0078 to 0.0184] | 0.0202 [0.0091 to 0.0446]
  Cycle 9 | 0.0161 [0.0114 to 0.0227] | 0.0153 [0.0105 to 0.0225] | 0.0202 [0.0091 to 0.0446]
  Cycle 10 | 0.0184 [0.0133 to 0.0255] | 0.0174 [0.0121 to 0.0250] | 0.0243 [0.0116 to 0.0507]
  Cycle 11 | 0.0190 [0.0138 to 0.0262] | 0.0181 [0.0127 to 0.0258] | 0.0243 [0.0116 to 0.0507]
  Cycle 12 | 0.0209 [0.0153 to 0.0284] | 0.0195 [0.0138 to 0.0276] | 0.0287 [0.0143 to 0.0570]
  Cycle 13 | 0.0247 [0.0185 to 0.0329] | 0.0240 [0.0175 to 0.0329] | 0.0287 [0.0143 to 0.0570]

5. Primary Outcome: Typical-Use Pregnancy Rates Based on Pearl Index (PI) Analyses for 28-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight, Using the 7-Day Rule
Description: Contraceptive failure is measured by the pregnancy rate calculated using the Pearl Index (PI) and the 7-day rule (a standardized process for calculating pregnancy rates). PI used all pregnancies, as determined by a positive urine and/or serum pregnancy test, except those for which the date of conception was before starting DR-102 or > 7 days after stopping the combination DSG/EE or EE treatment of DR-102.The PI is defined as number of contraceptive failures per 100 women-years of exposure: (100)*(total number of pregnancies)*(13)/(total number of 28-day cycles). Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'Typical-use' set included PITT participants who completed at least one 28-day cycle and in which no other birth control method (BCM), including condoms, were used.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Units Other Than Participants: Treatment Cycles
Arm/Group | DR-102: Total | DR-102: Baseline Body Weight <90 kg | DR-102: Baseline Body Weight ≥90 kg
Number analyzed (Participants) | 2333 | 1977 | 356
Number analyzed (Treatment Cycles) | 22309 | 19086 | 3223
pregnancies / 100 woman years exposure | 2.68 [1.963 to 3.574] | 2.59 [1.832 to 3.551] | 3.23 [1.394 to 6.350]

6. Primary Outcome: Compliant-Use Pregnancy Rates Based on Pearl Index (PI) Analyses for 28-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight, Using the 7-Day Rule
Description: Contraceptive failure is measured by the pregnancy rate calculated using the Pearl Index (PI) and the 7-day rule (a standardized process for calculating pregnancy rates). PI used all pregnancies, as determined by a positive urine and/or serum pregnancy test, except those for which the date of conception was before starting DR-102 or > 7 days after stopping the combination DSG/EE or EE treatment of DR-102.The PI is defined as number of contraceptive failures per 100 women-years of exposure: (100)*(total number of pregnancies)*(13)/(total number of 28-day cycles). Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets. Compliant use: did not skip 2 or more consecutive pills, had an overall compliance with IP administration of at least 80%, and did not use a prohibited medication.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. 'Compliant-use' set included PITT participants who completed at least one 28-day cycle and in which no other birth control method (BCM), including condoms, were used, and who were deemed to be compliant, per protocol.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Units Other Than Participants: Treatment Cycles
Arm/Group | DR-102: Total | DR-102: Baseline Body Weight <90 kg | DR-102: Baseline Body Weight ≥90 kg
Number analyzed (Participants) | 2317 | 1961 | 356
Number analyzed (Treatment Cycles) | 22085 | 18886 | 3199
pregnancies / 100 woman years exposure | 2.00 [1.386 to 2.796] | 1.79 [1.169 to 2.621] | 3.25 [1.404 to 6.398]

7. Secondary Outcome: Compliant-Use Life-Table Estimates of Pregnancy Rates Based on 28-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: A life table approach was used to estimate the cumulative pregnancy rate on a cycle-by-cycle basis for each of the thirteen 28-day treatment cycles. Compliant use: did not skip 2 or more consecutive pills, had an overall compliance with IP administration of at least 80%, and did not use a prohibited medication.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'Compliant-use' set included PITT participants who completed at least one 28-day cycle and in which no other BCMs, including condoms, were used, and who were deemed to be compliant, per protocol.
Measure: Number (95% Confidence Interval); unit: pregnancies / cumulative exposure
Arm/Group | DR-102: Total | DR-102: Baseline Body Weight <90 kg | DR-102: Baseline Body Weight ≥90 kg
Number analyzed (Participants) | 2317 | 1961 | 356
pregnancies / cumulative exposure
  Cycle 1 | 0 [0.0000 to 0.0000] | 0 [0.0000 to 0.0000] | 0 [0.0000 to 0.0000]
  Cycle 2 | 0.0015 [0.0004 to 0.0059] | 0.0009 [0.0001 to 0.0062] | 0.0047 [0.0007 to 0.0330]
  Cycle 3 | 0.0038 [0.0016 to 0.0092] | 0.0037 [0.0014 to 0.0098] | 0.0047 [0.0007 to 0.0330]
  Cycle 4 | 0.0063 [0.0032 to 0.0126] | 0.0046 [0.0019 to 0.0111] | 0.0154 [0.0050 to 0.0472]
  Cycle 5 | 0.0063 [0.0032 to 0.0126] | 0.0046 [0.0019 to 0.0111] | 0.0154 [0.0050 to 0.0472]
  Cycle 6 | 0.0063 [0.0032 to 0.0126] | 0.0046 [0.0019 to 0.0111] | 0.0154 [0.0050 to 0.0472]
  Cycle 7 | 0.0072 [0.0038 to 0.0139] | 0.0057 [0.0026 to 0.0128] | 0.0154 [0.0050 to 0.0472]
  Cycle 8 | 0.0102 [0.0058 to 0.0179] | 0.0080 [0.0040 to 0.0160] | 0.0224 [0.0084 to 0.0593]
  Cycle 9 | 0.0152 [0.0095 to 0.0245] | 0.0139 [0.0081 to 0.0239] | 0.0224 [0.0084 to 0.0593]
  Cycle 10 | 0.0163 [0.0103 to 0.0258] | 0.0139 [0.0081 to 0.0239] | 0.0298 [0.0124 to 0.0712]
  Cycle 11 | 0.0163 [0.0103 to 0.0258] | 0.0139 [0.0081 to 0.0239] | 0.0298 [0.0124 to 0.0712]
  Cycle 12 | 0.0174 [0.0111 to 0.0272] | 0.0152 [0.0090 to 0.0256] | 0.0298 [0.0124 to 0.0712]
  Cycle 13 | 0.0208 [0.0137 to 0.0315] | 0.0191 [0.0119 to 0.0307] | 0.0298 [0.0124 to 0.0712]

8. Secondary Outcome: Percentage of On-Drug Pregnancies in All Users, by Body Weight Decile Groups Using the 7-Day Rule
Description: Crude pregnancy rate is defined as the percentage of on-drug pregnancies per number of participants in each body weight decile (weight range, in kilograms). The 7-day rule is a standardized process for calculating pregnancy rates. Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'All Users' set included PITT participants who completed at least one 28-day cycle. n=number of participants in the body weight decile group.
Measure: Number; unit: percentage of pregnancies
Arm/Group | DR-102
Number analyzed (Participants) | 2401
percentage of pregnancies
  ≤53.1 kg (n=249) | 0.40
  >53.1 to ≤57.1 kg (n=248) | 2.42
  >57.1 to ≤60.8 kg (n=249) | 1.61
  >60.8 to ≤64.0 kg (n=234) | 1.28
  >64.0 to ≤67.6 kg (n=222) | 4.05
  >67.6 to ≤72.1 kg (n=249) | 1.20
  >72.1 to ≤77.4 kg (n=230) | 2.17
  >77.4 to ≤85.3 kg (n=251) | 1.99
  >85.3 to ≤97.5 kg (n=236) | 2.12
  >97.5 to ≤181.4 kg (n=233) | 2.15

9. Secondary Outcome: Percentage of On-Drug Pregnancies in Typical-Use, by Body Weight Decile Groups Using the 7-Day Rule
Description: as for outcome 8
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'Typical-use' set included PITT participants who completed at least one 28-day cycle and in which no other birth control method (BCM), including condoms, were used. n=number of participants in body weight decile group.
Measure: Number; unit: percentage of pregnancies
Arm/Group | DR-102
Number analyzed (Participants) | 2333
percentage of pregnancies
  ≤53.1 kg (n=240) | 0.42
  >53.1 to ≤57.1 kg (n=240) | 2.50
  >57.1 to ≤60.8 kg (n=245) | 1.63
  >60.8 to ≤64.0 kg (n=227) | 1.32
  >64.0 to ≤67.6 kg (n=217) | 4.15
  >67.6 to ≤72.1 kg (n=240) | 1.25
  >72.1 to ≤77.5 kg (n=226) | 2.21
  >77.5 to ≤85.3 kg (n=242) | 2.07
  >85.3 to ≤97.1 kg (n=223) | 2.24
  >97.1 to ≤181.4 kg (n=233) | 2.15

10. Secondary Outcome: Percentage of On-Drug Pregnancies in Compliant-Use, by Body Weight Decile Groups Using the 7-Day Rule
Description: Crude pregnancy rate is defined as the percentage of on-drug pregnancies per number of participants in each body weight decile (weight range, in kilograms). The 7-day rule is a standardized process for calculating pregnancy rates. Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets. Compliant use: did not skip 2 or more consecutive pills, had an overall compliance with IP administration of at least 80%, and did not use a prohibited medication.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. 'Compliant-use' set included PITT participants who completed at least 1 28-day cycle in which no other BCMs were used, and who were deemed to be compliant, per protocol. n=number of participants in body weight decile group.
Measure: Number; unit: percentage of pregnancies
Arm/Group | DR-102
Number analyzed (Participants) | 2317
percentage of pregnancies
  ≤53.1 kg (n=238) | 0.42
  >53.1 to ≤57.1 kg (n=240) | 1.67
  >57.1 to ≤60.8 kg (n=244) | 1.23
  >60.8 to ≤64.0 kg (n=225) | 0.89
  >64.0 to ≤67.6 kg (n=215) | 2.79
  >67.6 to ≤72.1 kg (n=237) | 0.84
  >72.1 to ≤77.5 kg (n=223) | 2.24
  >77.5 to ≤85.3 kg (n=241) | 0.83
  >85.3 to ≤97.5 kg (n=228) | 1.75
  >97.5 to ≤181.4 kg (n=226) | 2.21

11. Secondary Outcome: Percentage of On-Drug Pregnancies in All Users, by Body Mass Index (BMI) Decile Groups Using the 7-Day Rule
Description: Crude pregnancy rate is defined as the percentage of on-drug pregnancies per number of participants in each body mass index (BMI) decile (BMI range, in kg/m^2). The 7-day rule is a standardized process for calculating pregnancy rates. Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'All Users' set included PITT participants who completed at least one 28-day cycle. n=number of participants in BMI decile group.
Measure: Number; unit: percentage of pregnancies
Arm/Group | DR-102
Number analyzed (Participants) | 2401
percentage of pregnancies
  ≤20.1 kg/m^2 (n=243) | 1.65
  >20.1 to ≤21.5 kg/m^2 (n=238) | 1.68
  >21.5 to ≤22.7 kg/m^2 (n=240) | 1.67
  >22.7 to ≤23.8 kg/m^2 (n=241) | 0.83
  >23.8 to ≤25.2 kg/m^2 (n=240) | 1.25
  >25.2 to ≤26.6 kg/m^2 (n=242) | 2.07
  >26.6 to ≤28.7 kg/m^2 (n=237) | 2.11
  >28.7 to ≤31.4 kg/m^2 (n=240) | 3.33
  >31.4 to ≤35.6 kg/m^2 (n=241) | 2.49
  >35.6 to ≤68.0 kg/m^2 (n=239) | 2.09

12. Secondary Outcome: Percentage of On-Drug Pregnancies in Typical-Use, by Body Mass Index (BMI) Decile Groups Using the 7-Day Rule
Description: as for outcome 11
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. The 'Typical-use' set included PITT participants who completed at least one 28-day cycle and in which no other birth control method (BCM), including condoms, were used. n=number of participants in BMI decile group.
Measure: Number; unit: percentage of pregnancies
Arm/Group | DR-102
Number analyzed (Participants) | 2333
percentage of pregnancies
  ≤20.1 kg/m^2 (n=235) | 1.70
  >20.1 to ≤21.5 kg/m^2 (n=233) | 1.72
  >21.5 to ≤22.7 kg/m^2 (n=232) | 1.72
  >22.7 to ≤23.8 kg/m^2 (n=235) | 0.85
  >23.8 to ≤25.2 kg/m^2 (n=232) | 1.29
  >25.2 to ≤26.6 kg/m^2 (n=233) | 2.15
  >26.6 to ≤28.7 kg/m^2 (n=234) | 2.14
  >28.7 to ≤31.4 kg/m^2 (n=233) | 3.43
  >31.4 to ≤35.7 kg/m^2 (n=233) | 2.58
  >35.7 to ≤68.0 kg/m^2 (n=233) | 2.15

13. Secondary Outcome: Percentage of On-Drug Pregnancies in Compliant-Use, by Body Mass Index (BMI) Decile Groups Using the 7-Day Rule
Description: Crude pregnancy rate is defined as the percentage of on-drug pregnancies per number of participants in each body mass index (BMI) decile (BMI range, in kg/m^2). The 7-day rule is a standardized process for calculating pregnancy rates. Seven-day rule: a pregnancy was considered "on drug" if the date of conception was on or after the date of first dose of investigational product (IP), but no more than 7 days after the last tablet was taken; last tablet included combination hormonal or EE tablets. Compliant use: did not skip 2 or more consecutive pills, had an overall compliance with IP administration of at least 80%, and did not use a prohibited medication.
Time Frame: thirteen 28-day cycles
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age, inclusive, at the Screening Visit. 'Compliant-use' set included PITT participants who completed at least 1 28-day cycle and in which no other BCMs were used, and who were deemed to be compliant, per protocol. n=number of participants in BMI decile group.
Measure: Number; unit: percentage of pregnancies
Arm/Group | DR-102
Number analyzed (Participants) | 2317
percentage of pregnancies
  ≤20.1 kg/m^2 (n=233) | 0.86
  >20.1 to ≤21.5 kg/m^2 (n=231) | 1.30
  >21.5 to ≤22.7 kg/m^2 (n=239) | 0.84
  >22.7 to ≤23.8 kg/m^2 (n=225) | 0.89
  >23.8 to ≤25.2 kg/m^2 (n=232) | 0.86
  >25.2 to ≤26.6 kg/m^2 (n=233) | 1.29
  >26.6 to ≤28.7 kg/m^2 (n=229) | 2.18
  >28.7 to ≤31.4 kg/m^2 (n=232) | 2.59
  >31.4 to ≤35.7 kg/m^2 (n=233) | 1.72
  >35.7 to ≤68.0 kg/m^2 (n=230) | 2.17

ADVERSE EVENTS:
Time Frame: Serious adverse Event (SAE) reporting period began upon signed informed consent and ended at the Final Study or the Early Withdrawal Visit. AEs were reported at each study visit (Weeks 0 through Week 53). Treatment duration with IP was up to one year.
Arm/Group | DR-102
Serious Adverse Events (participants affected / at risk) | 46/2765
Other Adverse Events (participants affected / at risk) | 1319/2765
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DR-102 (N=2765)
Anaemia (Blood and lymphatic system disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Biliary dyskinesia (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Meningitis viral (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Toxic shock syndrome streptococcal (Infections and infestations) | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1
Alpha 1 foetoprotein increased (Investigations) | 1
Foetal heart rate decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Narcolepsy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 5
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Panic disorder with agoraphobia (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 2
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DR-102 (N=2765)
Nausea (Gastrointestinal disorders) | 130
Vomiting (Gastrointestinal disorders) | 47
Nasopharyngitis (Infections and infestations) | 247
Upper respiratory infection (Infections and infestations) | 172
Sinusitus (Infections and infestations) | 152
Urinary tract infection (Infections and infestations) | 130
Vulvovaginal mycotic infection (Infections and infestations) | 128
Vaginitis bacterial (Infections and infestations) | 105
Bronchitis (Infections and infestations) | 67
Pharyngitis streptococcal (Infections and infestations) | 55
Gastroenteritis viral (Infections and infestations) | 53
Influenza (Infections and infestations) | 42
Weight increased (Investigations) | 108
Human papilloma virus test positive (Investigations) | 43
Headache (Nervous system disorders) | 132
Migraine (Nervous system disorders) | 51
Anxiety (Psychiatric disorders) | 54
Depression (Psychiatric disorders) | 43
Metrorrhagia (Reproductive system and breast disorders) | 121
Cervical dysplasia (Reproductive system and breast disorders) | 114
Dysmenorrhea (Reproductive system and breast disorders) | 82
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 46
Acne (Skin and subcutaneous tissue disorders) | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/Institution must submit proposed publication to Sponsor for review within a prespecified number of days before submission for publication. If Sponsor's review shows that potentially patentable subject matter would be disclosed, publication/public disclosure shall be delayed to enable Sponsor, or Sponsor's designees, to file necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.